CLINICAL TRIAL: NCT05838664
Title: SIFNOS STUDY: RETROSPECTIVE STUDY IN PATIENTS WITH ATRIAL FIBRILLATION (AF) EXPOSED AND UNEXPOSED TO AN ORAL ANTICOAGULANT THERAPY BETWEEN 2016-2020 IN FRANCE
Brief Title: A Study to Learn About the Effects of Medicines That Help in Thinning the Blood in People With Atrial Fibrillation (AF) Between 2016 and 2020 in France
Acronym: SIFNOS
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B0661173; SIFNOS (Other: Alias Study Number)
Record Dates: First submitted 2023-03-28; First posted 2023-05-01 (Actual); Results first posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation | interventions — apixaban; Rivaroxaban; Dabigatran

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (5):
- AF patients unexposed to oral anticoagulants
  Interventions: Drug: No OAC
- AF patients exposed to VKA
  Interventions: Drug: VKA
- AF patients exposed to apixaban
  Interventions: Drug: apixaban
- AF patients exposed to rivaroxaban
  Interventions: Drug: rivaroxaban
- AF patients exposed to dabigatran
  Interventions: Drug: dabigatran

INTERVENTIONS:
Drug: No OAC — AF Patient who were not exposed to oral anticoagulation
  Groups: AF patients unexposed to oral anticoagulants
Drug: VKA — AF patients who received VKA
  Groups: AF patients exposed to VKA
Drug: apixaban — AF patients who received apixaban
  Groups: AF patients exposed to apixaban
Drug: rivaroxaban — AF patients who received rivaroxaban
  Groups: AF patients exposed to rivaroxaban
Drug: dabigatran — AF patients who received dabigatran
  Groups: AF patients exposed to dabigatran

SUMMARY:
The purpose of this study is to look at how many patients with AF had strokes, major bleeding and death in both people who had and had not taken any oral anticoagulant. Atrial fibrillation (AF) is an irregular and often very rapid heart rhythm (arrhythmia) that can lead to blood clots in the heart.

This increases the risk of stroke. Anticoagulants are medicines, also called blood thinners, which help prevent blood clots from forming or getting bigger.

This study includes patient's data from the database who:

* Had at least one hospital stay with AF
* Are new users of OACs for AF treatment
* Are 18 years and older when they were confirmed to have AF All the patient's data included in this study would have either received the OAC therapy or not.

This study aims to look at any events of strokes, major bleeding and death. The data of patients will be collected from the French national health insurance claims database (SNDS). The planned study period is thought to be from 1st January 2016 till 31st December 2020

ELIGIBILITY:
Inclusion Criteria:

* Identified patients with AF aged 18 years and older at diagnosis of AF

Exclusion Criteria:

* AF Patients with at least one hospital stays for associated valve disease or valve surgery
* Patients treated with an OAC for another indication than AF

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 18 years old AF Patients and older will be included from January 1st, 2016 to December 31st, 2020:
Sampling Method: Non-Probability Sample
Enrollment: 2140403 (Actual)
Dates: Start 2023-07-07 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer Investigational Site, Paris, France

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B0661173

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Retrospective data on eligible atrial fibrillation (AF) participants were collected from French National Health Data System (Systeme National des Donnees de Sante) (01-Jan-2016 and 31-Dec-2019; maximum up to 48 months), with a 2-year historical period before index date; study conducted in France. Available data was evaluated as per study objectives, from 07-Jul-2023 to 30-Sep-2024 (approximately 14 months) in this retrospective observational study.
Groups:
- Participants Exposed to OACs: Participants with AF who were exposed to vitamin K antagonist (VKA) or direct oral anticoagulant ([DOACs] including apixaban, rivaroxaban or dabigatran) and were identified from Systeme National des Donnees de Sante (SNDS) databases between 01-Jan-2016 and 31-Dec-2019, with a 2-year historical period before index date were included.
- Participants Unexposed to OACs: Participants with AF who were unexposed to VKA or DOACs including apixaban, rivaroxaban or dabigatran) and were identified from SNDS databases between 01-Jan-2016 and 31-Dec-2019, with a 2-year historical period before index date were included.
Period: Overall Study
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Started | 1583444 | 556959
Completed | 1583444 | 556959
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were analyzed in the Incident AF population which was defined as participants newly diagnosed with AF (i.e. no AF diagnostic during the historical period) from 01-Jan-2016 to 31-Dec-2019 (inclusion period).
Groups:
- Participants Exposed to OACs: Participants with AF who were exposed to VKA or DOACs (including apixaban, rivaroxaban or dabigatran) within 30 days after inclusion and were identified from SNDS databases between 01-Jan-2016 and 31-Dec-2019 were included.
- Participants Unexposed to OACs: Participants with AF who were unexposed to OACs within 30 days after inclusion and were identified from SNDS between 01-Jan-2016 and 31-Dec-2019 were included.
- Total: Total of all reporting groups
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs | Total
Number analyzed (Participants) | 943648 | 446645 | 1390293
Age, Customized [Count of Participants; unit: Participants]
  <80 years | 528010 | 212865 | 740875
  80-90 years | 321396 | 149231 | 470627
  >=90 years | 94242 | 84549 | 178791
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 415404 | 219829 | 635233
  Male | 528244 | 226816 | 755060
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Incidence Rate (Per 1000 Participant-years) of Stroke in Non-valvular Atrial Fibrillation (AF) Participants Exposed to Oral Anticoagulation (OAC) and Unexposed to OAC
Description: Incidence rate was defined as the number of events occurring during the follow-up period divided by the number of person-years of follow-up (sum of durations of follow-up period for incident participants). Incidence rate of stroke (ischemic or hemorrhage) in non-valvular AF participants who were exposed to OAC or unexposed to OAC were reported in this outcome measure. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: Follow up period: From index date until death, end of study or the date of last reimbursement of care recorded in the SNDS (maximum up to 48 months); retrospective data was retrieved and analyzed during approximately 9 months of this observational study
Population: Certain AF incident population included participants with a first AF diagnosis date during study period but without history of OACs delivery in the 24 months before inclusion date, with no reported events of interest (stroke, major bleeding) between inclusion and index date. Here, ''Overall number of participants analyzed'' signifies participants evaluable for this outcome measure.
Measure: Number (95% Confidence Interval); unit: Events per 1000 person years
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 556876 | 505597
Events per 1000 person years | 14.7 [14.4 to 15.0] | 31.2 [30.7 to 31.6]

2. Primary Outcome: Incidence Rate (Per 1000 Participant-years) of Major Bleeding in Non-valvular AF Participants Exposed to OAC and Unexposed to OAC
Description: Incidence rate was defined as the number of events occurring during the follow-up period divided by the number of person-years of follow-up (sum of durations of follow-up period for incident participants). Incidence rate of major bleeding in non-valvular AF participants who were exposed to OAC or unexposed to OAC were reported in this outcome measure. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 person years
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 560862 | 503300
Events per 1000 person years | 21.5 [21.2 to 21.9] | 23.6 [23.2 to 24.0]

3. Primary Outcome: Incidence Rate (Per 1000 Participant-years) of Death in Non-valvular AF Participants Exposed to OAC and Unexposed to OAC
Description: Incidence rate was defined as the number of events occurring during the follow-up period divided by the number of person-years of follow-up (sum of durations of follow-up period for incident participants). Incidence rate of death in non-valvular AF participants who were exposed to OAC or unexposed to OAC were reported in this outcome measure. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Events per 1000 person years
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 562241 | 509072
Events per 1000 person years | 41.1 [40.7 to 41.6] | 184.6 [183.6 to 185.7]

4. Primary Outcome: Number of Participants With Contraindications to OAC at Index Date in Non-valvular AF Participants Exposed to OAC and Unexposed to OAC
Description: Contraindications included end-stage renal disease on dialysis, diseases of the blood and blood-forming organs, certain disorders involving the immune mechanism, recent history of acute bleeding gastric or duodenal ulcer, hepatic cirrhosis or fibrosis or liver failure. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: At index date (anytime in between 01-Jan-2016 and 31-Dec-2019); retrospective data was retrieved and analyzed during approximately 9 months of this observational study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Participants | 49478 | 86646

5. Primary Outcome: Number of Participants Who Received Complimentary Universal Health Care (CMU-c) in Non-valvular AF Participants Exposed to OAC and Unexposed to OAC
Description: A participant was considered to have received CMU-c if the participant benefitted from an exemption from care on the grounds of CMU-c for care received on the index date. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Participants | 12819 | 10198

6. Primary Outcome: Number of Participants Who Received Aid for Complementary Health Care (ACS) for Elderly Participants in Non-valvular AF Participants Exposed to OAC and Unexposed to OAC
Description: A participant was considered to have received ACS if the participant benefitted from an aid for complementary health care on the index date. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Participants | 10444 | 8698

7. Primary Outcome: Number of Participants Classified as Per Area of Residence in Non-valvular AF Participants Exposed to OAC and Unexposed to OAC
Description: Area of residence was derived based on the code of the department of residence recorded with health cares carried out on index date. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Participants
  Auvergne-Rhône-Alpes | 56168 | 34422
  Bourgogne-Franche-Comté | 24185 | 13849
  Bretagne | 25892 | 15574
  Centre-Val de Loire | 19626 | 14146
  Corse | 2689 | 1829
  Overseas districts and territories | 281 | 135
  Grand-Est | 43950 | 30014
  Hauts-de-France | 44740 | 30567
  Ile de France | 62389 | 45815
  Normandie | 26059 | 16507
  Nouvelle Aquitaine | 51529 | 33123
  Occitanie | 47963 | 30580
  Pays de la Loire | 25684 | 16155
  Provence-Alpes-Côte d Azur | 42929 | 28422
  Unknown | 11562 | 21098

8. Primary Outcome: Number of Participants Classified as Per Modified CHA2DS2-VASc Score in Non-valvular AF Participants Exposed to OAC and Unexposed to OAC
Description: Congestive heart failure, hypertension, age (>65 = 1 point, >75 = 2 points), diabetes, previous stroke/transient ischemic attack (2 points) (CHA2DS2)-vascular disease and sex category (VASc) scoring scale was used to estimate the risk of stroke and systemic emboli in participants with NVAF. CHA2DS2-VASc score was calculated based on 8 risk factors (age 65-74 years, age >=75 years, sex category, congestive heart failure history, hypertension history, stroke/transient ischemic attack/thromboembolism history, vascular disease history and diabetes mellitus history). Total CHA2DS2-VASc score ranged from 0-9 where 0= low risk and 9= high risk of stroke, higher scores indicated higher risk of stroke and systemic emboli. Index date was date of first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Participants
  High | 402191 | 281168
  Moderate | 57481 | 30413
  Low | 25974 | 20655

9. Primary Outcome: HAS-BLED Score in Non-valvular AF Participants Exposed to OAC and Unexposed to OAC
Description: HAS-BLED scoring scale was used to estimate the risk of bleeding. HAS-BLED score was calculated based on 9 risk factors (hypertension, renal disease, liver disease, stroke history, prior major bleeding or predisposition to bleeding, labile international normalized ratio (INR), age >65 years, medication usage predisposing to bleeding and alcohol use). Total HAS-BLED score ranged from 0 to 9 where 0 = low risk and >=3 = high risk of bleed, higher scores indicated more risk of bleeds. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Units on a scale | 2.26 (0.99) | 2.5 (1.10)

10. Primary Outcome: Number of Participants Classified as Per Type of Stroke in Non-valvular AF Participants Exposed to OAC and Unexposed to OAC
Description: Type of stroke was considered "Yes" if the participant was hospitalized with any discharge diagnosis (i.e., main and related diagnosis) of stroke (ischemic or hemorrhagic). Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 38623 | 48252
Participants
  Both Ischemic and haemorrhagic | 1285 | 5614
  Hemorrhagic | 1025 | 3996
  Ischemic | 36313 | 38642

11. Primary Outcome: Number of Participants With Risk of Falls in Non-valvular AF Participants Exposed to OAC and Unexposed to OAC
Description: Participants at risk of falls were identified by an algorithm adapted to SNDS data. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Participants | 186288 | 170465

12. Primary Outcome: Number of Participants Who Were Polymedicated in Non-valvular AF Participants Exposed to OAC and Unexposed to OAC
Description: Participant was considered polymedicated if the participant had reimbursements for greater than or equal to (>=) 5 different medications (different Anatomical Therapeutic Chemical codes [ATC] in the year before the index date. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: Up to 1 year prior to index date (index date was anytime in between 01-Jan-2016 and 31-Dec-2019); retrospective data was retrieved and analyzed during approximately 9 months of this observational study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Participants | 408403 | 291508

13. Primary Outcome: Number of Participants With Atleast One Visit to Nursing Home in Non-valvular AF Participants Exposed to OAC and Unexposed to OAC
Description: Participant was considered to have at least one visit to nursing home if the participant had at least one reimbursement corresponding to a nursing home on or in the 2 years prior to the index date. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: Up to 2 years prior to index date (index date was anytime in between 01-Jan-2016 and 31-Dec-2019); retrospective data was retrieved and analyzed during approximately 9 months of this observational study
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Participants | 16170 | 31493

14. Primary Outcome: Age Adjusted Charlson Comorbidity Index (CCI) in Non-valvular AF Participants Exposed to OAC and Unexposed to OAC
Description: CCI based on various comorbid conditions such as myocardial infarction, congestive heart failure (CHF), peripheral vascular disease, cerebrovascular disease, dementia, chronic obstructive pulmonary disease, rheumatologic disease, peptic ulcer disease, mild liver disease, diabetes (mild to moderate), diabetes + complications, hemiplegia or paraplegia, renal disease, any malignancy (lymphoma and leukemia), moderate/severe liver disease, metastatic solid tumor, and acquired immune deficiency syndrome (AIDS) were reported. The comorbidities were assessed with different weights (from 1 to 6), and the total score was determined by adding the scores of each comorbidity. CCI score range was from 0 to 14, where 0= low comorbid condition and 14= high comorbid condition, higher scores= more comorbidity. Index date = date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Units on a scale | 2.32 (2.06) | 3.6 (3.51)

15. Primary Outcome: Number of Participants Classified as Per Comorbidities in Non-valvular AF Participants Who Were Exposed to OAC and Unexposed to OAC
Description: The number of participants classified as per comorbidities (coronary arterial diseases, vascular and neurodegenerative dementia, myocardial infarction, congestive heart failure, peripheral arterial disease, other vascular diseases, sleep disorders, active cancer, malnutrition, morbid obesity, anemia, chronic obstructive pulmonary disease, diabetes, diabetes with complication, connective tissue disease, ulcer disease, cerebrovascular disease, cerebrovascular disease, mild liver disease, moderate-to-severe liver disease, hemiplegia) in non-valvular AF participants who were exposed to OAC and unexposed to OAC were reported in this outcome measure. One participant could have more than one comorbidity. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Participants
  Coronary arterial diseases | 86531 | 75022
  Vascular and neurodegenerative dementia | 23398 | 46852
  Myocardial infarction | 12063 | 8689
  Congestive heart failure | 87559 | 75117
  Peripheral arterial disease | 24219 | 30313
  Other vascular diseases | 7843 | 10216
  Sleep disorders | 18149 | 16376
  Active cancer | 75261 | 86281
  Malnutrition | 34650 | 78027
  Morbid obesity | 41052 | 34823
  Anemia | 14756 | 30332
  Chronic obstructive pulmonary disease | 2654 | 3942
  Diabetes | 99628 | 67412
  Diabetes with complication | 1165 | 1322
  Connective tissue disease | 8376 | 6960
  Ulcer disease | 2691 | 6211
  Cerebrovascular disease | 48715 | 58186
  Moderate-to-severe renal disease | 29846 | 42083
  Mild liver disease | 7183 | 10801
  Moderate-to-severe liver disease | 1551 | 4234
  Hemiplegia | 4761 | 8159

16. Secondary Outcome: Number of Participants With Concomitant Treatments in Non-valvular AF Participants Who Were Exposed to OAC and Unexposed to OAC
Description: Concomitant treatments included beta-blockers, antihypertensives, antiplatelet drugs, other anticoagulants(heparin, other antithrombotic agents, direct thrombin inhibitors[except dabigatran]),non-steroidal anti-inflammatory drugs(NSAIDs), oral corticoids, proton pump inhibitors, selective serotonin reuptake inhibitor antidepressants(SSRIs),systemic azole antifungals, other cytochrome P(CYP) P450 3A4 inhibitors(ticagrelor, diltiazem, verapamil, amiodarone, macrolide [except spiramycine]),medical procedure of cardioversion, digitalis glycosides, nitrates derivatives, benzodiazepines, lipid-lowering drugs, glucose-lowering drugs, antiarrhythmics. One participant could receive more than one concomitant treatment. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 4
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Participants
  Beta-blockers | 330710 | 124236
  Antihypertensives | 354602 | 198727
  Antiplatelet drugs | 206611 | 150062
  Other anticoagulants | 30265 | 32487
  NSAIDs | 69466 | 40497
  Oral corticoids | 73061 | 52102
  Proton pump inhibitors | 215924 | 143103
  SSRIs | 37035 | 32378
  Systemic azole antifungals | 3104 | 3948
  Protease inhibitors | 109 | 97
  Other CYP P450 3A4 inhibitors | 190900 | 55864
  Medical procedure of cardioversion | 6317 | 2603
  Antiarrhythmics | 204717 | 61093
  Glucose-lowering drugs | 91864 | 54691
  Lipid-lowering drugs | 195863 | 104804
  Digitalis glycosides | 20783 | 5392
  Nitrate derivatives | 23082 | 17315
  Benzodiazepines | 127625 | 97568

17. Secondary Outcome: Annual Incidence Rate of Non-valvular AF in Participants Exposed to OAC and Unexposed to OAC
Description: Annual incidence rate of AF was calculated as the number of newly diagnosed non-valvular AF incidents to the number of inhabitants aged >=18 years in France at risk of AF, in the corresponding year. Incidence rate of AF according to the corresponding year is reported in this outcome measure. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: Anytime in 2016, 2017, 2018 and 2019; retrospective data was retrieved and analyzed during approximately 9 months of this observational study
Population: All AF incident participants included participants with/without OAC treatments before the index date. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: New cases per 1000 persons
Groups:
- Participants Exposed to OACs: Participants with AF who were exposed to VKA or DOACs including apixaban, rivaroxaban or dabigatran) and were identified from SNDS databases between 01-Jan-2016 and 31-Dec-2019, with a 2-year historical period before index date were included.
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 224490 | 91946
New cases per 1000 persons
  2016 | 4.31 [4.29 to 4.33] | 1.75 [1.74 to 1.76]
  2017: number analyzed (Participants) | 215505 | 83785
  2017 | 4.13 [4.12 to 4.15] | 1.59 [1.58 to 1.6]
  2018: number analyzed (Participants) | 202038 | 72872
  2018 | 3.86 [3.85 to 3.88] | 1.38 [1.37 to 1.39]
  2019: number analyzed (Participants) | 195852 | 64627
  2019 | 3.73 [3.71 to 3.74] | 1.22 [1.21 to 1.23]

18. Secondary Outcome: Annual Prevalence (Prevalent Cases Per 1000 Years) of Non-valvular AF in Participants Exposed to OAC and Unexposed to OAC
Description: Annual prevalence of non-valvular AF was defined as the number of diagnosed non-valvular atrial fibrillation (NVAF) participants to the number of inhabitants aged >=18 years in France, in the corresponding year (National Institute for Statistics and Economic Studies [INSEE] data). Prevalence of AF according to the corresponding year is reported in this outcome measure. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 17
Population: Prevalent AF participants included participants diagnosed with AF during the historical period of two years before the index date. Here, "Overall Number of Participants Analyzed" signifies number of participants evaluable for this outcome measure. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Number (95% Confidence Interval); unit: Prevalent cases per 1000 years
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 1141152 | 438600
Prevalent cases per 1000 years
  2016: number analyzed (Participants) | 788170 | 278376
  2016 | 1.50 [1.49 to 1.5] | 0.53 [0.53 to 0.53]
  2017: number analyzed (Participants) | 932652 | 345579
  2017 | 1.76 [1.76 to 1.77] | 0.65 [0.65 to 0.66]
  2018: number analyzed (Participants) | 1044991 | 396207
  2018 | 1.97 [1.96 to 1.97] | 0.75 [0.74 to 0.75]
  2019 | 2.13 [2.13 to 2.14] | 0.82 [0.82 to 0.82]

19. Secondary Outcome: Number of Participants Who Were New Users of OAC and VKA
Description: Participants were considered as new users of OAC and VKA if the participant received at least one reimbursement of an OAC (VKA, apixaban, rivaroxaban or dabigatran) during the inclusion period, without use of any OAC in the 24 months prior to the first date of OAC delivery. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 4
Population: Certain AF incident population included participants with a first AF diagnosis date during study period but without history of OACs delivery in the 24 months before inclusion date, with no reported events of interest (stroke, major bleeding) between inclusion and index date. Here, ''Overall number of participants analyzed (N)'' signifies participants evaluable for this outcome measure.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 601998 | 395461
Participants | 421313 | 0

20. Secondary Outcome: Number of Participants According to Number of Treatment Sequence
Description: Number of participants according to number of treatment sequence (only one sequence of treatment, at least two sequences of treatment) is reported in this outcome measure. Index date was the date of the first dispensation of OAC for participants exposed to OAC.
Time Frame: as for outcome 1
Population: Certain AF incident population included participants with a first AF diagnosis date during study period but without history of OACs delivery in the 24 months before inclusion date, with no reported events of interest (stroke, major bleeding) between inclusion and index date. Here, "N"=participants evaluable for this outcome measure who received at least one sequence of treatment. As pre-specified in protocol this outcome measure was planned to be analyzed only in participants exposed to OACs.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Exposed to OACs
Number analyzed (Participants) | 572290
Participants
  Only one sequence of treatment | 451539
  At least two sequences of treatment | 120751

21. Secondary Outcome: Duration of Each Sequence of OAC Treatment
Description: Duration of each sequence of OAC treatment (i.e., at least one sequence of OAC treatment and at least two sequences of OAC treatment) for the participants who were exposed to OAC were reported in this outcome measure. Index date was the date of the first dispensation of OAC for participants exposed to OAC.
Time Frame: as for outcome 1
Population: Certain AF incident population included participants with a first AF diagnosis date during study period but without history of OACs delivery in the 24 months before inclusion date, with no reported events of interest (stroke, major bleeding) between inclusion and index date. Here, "N"= participants evaluable for this outcome measure who received at least one sequence of treatment. As pre-specified in protocol this outcome measure was planned to be analyzed only in participants exposed to OACs.
Measure: Median (Full Range); unit: Months
Arm/Group | Participants Exposed to OACs
Number analyzed (Participants) | 572290
Months
  At least one sequence of treatment | 9.5 [2.8 to 22.3]
  At least two sequences of treatment: number analyzed (Participants) | 120751
  At least two sequences of treatment | 6.9 [2.4 to 15.5]

22. Secondary Outcome: Number of Participants With Treatment Switch of OAC Treatment
Description: The number of participants with treatment switch who were exposed to OAC were reported in this outcome measure. Treatment switch was categorized into following categories: at least one sequence of treatment and at least two sequences of treatment. At least one sequence of treatment was defined as one or more OAC was given, and at least two sequences of treatment was defined as two or more OACs were given. Participants were considered to have treatment switch if the participant had at least one reimbursement of a OAC different from the first OAC delivered. Index date was the date of the first dispensation of OAC for participants exposed to OAC.
Time Frame: as for outcome 1
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Exposed to OACs
Number analyzed (Participants) | 572290
Participants
  At least one sequence of treatment | 48101
  At least two sequences of treatment: number analyzed (Participants) | 120751
  At least two sequences of treatment | 8592

23. Secondary Outcome: Number of Participants With Temporary or Permanent Treatment Discontinuation of OAC
Description: Participants were considered to have temporary or permanent discontinuation if the participant had at least 60 days without reimbursement of an OAC after the date of the first OAC delivery. The number of participants with temporary or permanent discontinuation of OAC who were exposed to OAC were reported in this outcome measure. Index date was the date of the first dispensation of OAC for participants exposed to OAC. At least one sequence of treatment was defined as one or more OAC was given, and at least two sequences of treatment was defined as two or more OACs were given.
Time Frame: as for outcome 1
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Exposed to OACs
Number analyzed (Participants) | 572290
Participants
  At least one sequence of treatment | 167099
  At least two sequences of treatment: number analyzed (Participants) | 120751
  At least two sequences of treatment | 40849

24. Secondary Outcome: Number of Participants Classified According to Type of OAC Delivery for Participants Exposed to OACs
Description: The number of participants classified according to type of OAC delivery (apixaban, rivaroxaban, VKA, dabigatran) who were exposed to OAC were reported in this outcome measure. Index date was the date of the first dispensation of OAC for participants exposed to OAC.
Time Frame: as for outcome 4
Population: Certain AF incident population included participants with a first AF diagnosis date during study period but without history of OACs delivery in the 24 months before inclusion date, with no reported events of interest (stroke, major bleeding) between inclusion and index date. Here, ''Overall number of participants analyzed'' signifies participants evaluable for this outcome measure. As pre-specified in protocol this outcome measure was planned to be analyzed only in participants exposed to OACs.
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Exposed to OACs
Number analyzed (Participants) | 485646
Participants
  Apixaban | 245094
  Rivaroxaban | 151288
  VKA | 56632
  Dabigatran | 32632

25. Secondary Outcome: Number of Participants According to Speciality of Prescriber for Participant Exposed to OAC
Description: Specialty of prescriber in participants who were exposed to OAC were reported in this outcome measure. Categories included hospital-based physician, generalist practitioners, city cardiologist, other and not specified. Index date was the date of the first dispensation of OAC for participants exposed to OAC. At least one sequence of treatment was defined as one or more OAC was given, and at least two sequences of treatment was defined as two or more OACs were given.
Time Frame: as for outcome 1
Population: as for outcome 21
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Exposed to OACs
Number analyzed (Participants) | 572290
Participants
  At least one sequence of treatment: Hospital-based physician | 222102
  At least one sequence of treatment: Generalist practitioners | 100629
  At least one sequence of treatment: City cardiologist | 134893
  At least one sequence of treatment: Other | 114252
  At least one sequence of treatment: Not specified | 414
  At least two sequences of treatment: number analyzed (Participants) | 120751
  At least two sequences of treatment: Hospital-based physician | 27905
  At least two sequences of treatment: Generalist practitioners | 49635
  At least two sequences of treatment: City cardiologist | 19714
  At least two sequences of treatment: Other | 23300
  At least two sequences of treatment: Not specified | 197

26. Secondary Outcome: Mean Number of Hospital Stays Per Participant Per Month Before the First Stroke From 6 to 12 Months
Description: Mean number of hospital stays with and without emergency visit per participant per month from 6 to 12 months before the first stroke who were exposed to OAC and unexposed to OAC were reported in this outcome measure.
Time Frame: From 6 to 12 months before the first stroke (anytime during 01-Jan-2016 and 31-Dec-2019); retrospective data was retrieved and analyzed during approximately 9 months of this observational study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hospital stays per participant per month
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Hospital stays per participant per month | 0.2 (0.96) | 0.2 (0.88)

27. Secondary Outcome: Mean Number of Outpatient Visits Per Participant Per Month Before the First Stroke From 6 to 12 Months
Description: Outpatient visits including physicians visits (private practice and home), paramedic visits in community setting, public hospital outpatient visits (management services organization [MSO] and rehabilitation care facilities) are reported. Mean number of outpatient visits per participant per month from 6 to 12 months before the first stroke who were exposed to OAC and unexposed to OAC were reported in this outcome measure.
Time Frame: as for outcome 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Visits per participant per month
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Visits per participant per month
  Physicians visits (private practice and home) | 1.1 (0.86) | 1.0 (0.87)
  Paramedic visits in community setting | 29.7 (38.63) | 20.3 (30.11)
  Public hospital outpatient visits (MSO and rehabilitation care facilities) | 0.2 (0.39) | 0.1 (0.32)

28. Secondary Outcome: Mean Number of Laboratory Tests Per Participant Per Month (PPPM) Before the First Stroke From 6 to 12 Months
Description: Mean number of laboratory tests per participant per month from 6 to 12 months before the first stroke who were exposed to OAC and unexposed to OAC were reported in this outcome measure.
Time Frame: as for outcome 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Laboratory tests PPPM
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Laboratory tests PPPM | 1.0 (1.42) | 0.5 (0.85)

29. Secondary Outcome: Mean Number of Medical Procedures Per Participant Per Month Before the First Stroke From 6 to 12 Months
Description: Mean number of medical procedures per participant per month from 6 to 12 months before the first stroke who were exposed to OAC and unexposed to OAC were reported in this outcome measure.
Time Frame: as for outcome 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Procedures per participant per month
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Procedures per participant per month | 0.5 (0.63) | 0.5 (0.68)

30. Secondary Outcome: Mean Number of Reimbursed Transports Per Participant Per Month Before the First Stroke From 6 to 12 Months
Description: Mean number of reimbursed transports per participant per month from 6 to 12 months before the first stroke who were exposed to OAC and unexposed to OAC were reported in this outcome measure.
Time Frame: as for outcome 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Transport per participant per month
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Transport per participant per month | 0.4 (0.99) | 0.3 (0.92)

31. Secondary Outcome: Mean Number of Drugs Dispensed Per Participant Per Month Before the First Stroke From 6 to 12 Months
Description: Mean number of drugs dispensed per participant per month from 6 to 12 months before the first stroke who were exposed to OAC and unexposed to OAC were reported in this outcome measure.
Time Frame: as for outcome 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Drugs dispensed PPPM
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Drugs dispensed PPPM | 11.6 (7.44) | 9.1 (7.72)

32. Secondary Outcome: Mean Number of Medical Devices Dispensed Per Participant Per Month Before the First Stroke From 6 to 12 Months
Description: Mean number of medical devices dispensed per participant per month from 6 to 12 months before the first stroke who were exposed to OAC and unexposed to OAC were reported in this outcome measure.
Time Frame: as for outcome 26
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Medical devices dispensed PPPM
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Medical devices dispensed PPPM | 0.8 (1.29) | 0.6 (1.11)

33. Secondary Outcome: Mean Number of Hospital Stays Per Participant Per Month After the First Stroke From 6 to 12 Months
Description: Mean number of hospital stays per participant per month from 6 to 12 months after the first stroke who were exposed to OAC and unexposed to OAC were reported in this outcome measure.
Time Frame: From 6 to 12 months after the first stroke (anytime during 01-Jan-2016 and 31-Dec-2019); retrospective data was retrieved and analyzed during approximately 9 months of this observational study
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Hospital stays per participant per month
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Hospital stays per participant per month | 0.2 (1.04) | 0.3 (1.64)

34. Secondary Outcome: Mean Number of Outpatient Visits Per Participant Per Month After the First Stroke From 6 to 12 Months
Description: Outpatient visits included physicians visits (private practice and home), paramedic visits in community setting and public hospital outpatient visits (MSO and rehabilitation care facilities). Mean number of outpatient visits per participant per month from 6 to 12 months after the first stroke who were exposed to OAC and unexposed to OAC were reported in this outcome measure.
Time Frame: as for outcome 33
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Visits per participant per month
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Visits per participant per month
  Physicians visits (private practice and home) | 1.0 (1.01) | 0.9 (1.18)
  Paramedic visits in community setting | 35.3 (44.24) | 29.4 (43.55)
  Public hospital outpatient visits (MSO and rehabilitation care facilities) | 0.2 (0.38) | 0.2 (0.40)

35. Secondary Outcome: Mean Number of Laboratory Tests Per Participant Per Month After the First Stroke From 6 to 12 Months
Description: Mean number of laboratory tests per participant per month from 6 to 12 months after the first stroke who were exposed to OAC and unexposed to OAC were reported in this outcome measure.
Time Frame: as for outcome 33
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Laboratory tests PPPM
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Laboratory tests PPPM | 0.9 (1.48) | 0.6 (1.21)

36. Secondary Outcome: Mean Number of Outpatient Medical Procedures Per Participant Per Month of HCRU After the First Stroke From 6 to 12 Months
Description: Mean number of outpatient medical procedures per participant per month from 6 to 12 months after the first stroke who were exposed to OAC and unexposed to OAC were reported in this outcome measure.
Time Frame: as for outcome 33
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Procedures per participant per month
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Procedures per participant per month | 0.5 (0.70) | 0.4 (0.73)

37. Secondary Outcome: Mean Number of Reimbursed Transports Per Participant Per Month of HCRU After the First Stroke From 6 to 12 Months
Description: Mean number of reimbursed transports per participant per month from 6 to 12 months after the first stroke who were exposed to OAC and unexposed to OAC were reported in this outcome measure.
Time Frame: as for outcome 33
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Transport per participant per month
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Transport per participant per month | 0.5 (1.20) | 0.6 (1.48)

38. Secondary Outcome: Mean Number of Drugs Dispensed Per Participant Per Month After the First Stroke From 6 to 12 Months
Description: Mean number of drugs dispensed per participant per month of HCRU from 6 to 12 months after the first stroke who were exposed to OAC and unexposed to OAC were reported in this outcome measure.
Time Frame: as for outcome 33
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Drugs dispensed PPPM
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Drugs dispensed PPPM | 11.9 (10.66) | 9.2 (10.43)

39. Secondary Outcome: Mean Number of Medical Devices Dispensed Per Participant Per Month After the First Stroke From 6 to 12 Months
Description: Mean number of medical devices dispensed per participant per month of HCRU from 6 to 12 months after the first stroke who were exposed to OAC and unexposed to OAC were reported in this outcome measure.
Time Frame: as for outcome 33
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Medical devices dispensed PPPM
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Medical devices dispensed PPPM | 1.0 (1.88) | 1.0 (1.97)

40. Secondary Outcome: Hospitalization Cost in Participants Exposed to and Unexposed to OAC
Description: Hospitalization cost (Euros per participant per month) in participants who were exposed to and unexposed to OAC were reported in this outcome measure. Cost equals to the value of cost (i.e. including reimbursed and non-reimbursed amounts) indicated in the data extraction and associated with the reimbursement. All cost was calculated per participant per month (PPPM). Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Euros per participant per month
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Euros per participant per month | 434.1 (1885.73) | 1318.5 (32665.57)

41. Secondary Outcome: Medical Procedures and Blood Examination Cost in Participants Exposed to and Unexposed to OAC
Description: Medical procedures and blood examination cost (Euros per participant per month) in participants who were exposed to and unexposed to OAC were reported in this outcome measure. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study. Certain AF incident population included participants with a first AF diagnosis date during study period but without history of OACs delivery in the 24 months before inclusion date, with no reported events of interest (stroke, major bleeding) between inclusion and index date.
Time Frame: as for outcome 1
Population: Certain AF incident population. Here, ''Overall number of participants analysed'' signifies participants evaluable for this outcome measure. All participants reported under 'N' contributed data to the table; however, may not have evaluable data for each row. Here, "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Euros per participant per month
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 413397 | 309834
Euros per participant per month
  Outpatient medical procedures (public and private settings): number analyzed (Participants) | 361232 | 221892
  Outpatient medical procedures (public and private settings) | 33.1 (101.54) | 28.2 (162.60)
  Blood examination: number analyzed (Participants) | 369569 | 214065
  Blood examination | 14.3 (24.54) | 11.2 (31.92)

42. Secondary Outcome: Mean Number of Hospital Stays Per Month
Description: Mean number of hospital stays per month for participants who were exposed to OAC and unexposed to OAC were reported in this outcome measure. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study. Certain AF incident population included participants with a first AF diagnosis date during study period but without history of OACs delivery in the 24 months before inclusion date, with no reported events of interest (stroke, major bleeding) between inclusion and index date.
Time Frame: as for outcome 1
Population: Certain AF incident population. Here, ''Overall number of participants analyzed'' signifies participants evaluable for this outcome measure and "Number Analyzed" signifies number of participants evaluable for specified rows.
Measure: Mean (Standard Deviation); unit: Hospital stays per month
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 183966 | 135673
Hospital stays per month
  MSO hospital stays with and without emergency visit (public and private settings) | 0.2 (1.00) | 0.4 (1.77)
  MSO hospital stays starting with emergency visit (public and private settings): number analyzed (Participants) | 79567 | 61627
  MSO hospital stays starting with emergency visit (public and private settings) | 0.0 (0.27) | 0.1 (0.46)
  Hospital stays in rehabilitation care facilities: number analyzed (Participants) | 20825 | 26586
  Hospital stays in rehabilitation care facilities | 0.0 (0.07) | 0.0 (0.52)
  MSO hospital stays with palliative care (public and private settings): number analyzed (Participants) | 4662 | 10007
  MSO hospital stays with palliative care (public and private settings) | 0.0 (0.08) | 0.0 (0.40)

43. Secondary Outcome: Mean Number of Emergency Visits Per Month
Description: Mean number of emergency visits per month for participants who were exposed to OAC and unexposed to OAC were reported in this outcome measure. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Emergency visits per month
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 72022 | 50666
Emergency visits per month | 0.0 (0.23) | 0.0 (0.20)

44. Secondary Outcome: Mean Number of Physician Visits
Description: Mean number of physician visits for participants who were exposed to OAC and unexposed to OAC were reported in this outcome measure. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Physician visits
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 400299 | 248409
Physician visits | 1.0 (1.08) | 0.8 (1.04)

45. Secondary Outcome: Mean Number of Public Hospital Outpatient Visits
Description: Mean number of public hospital outpatient visits for participants who were exposed to OAC and unexposed to OAC were reported in this outcome measure. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Outpatient visits
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 195674 | 132843
Outpatient visits | 0.2 (0.44) | 0.2 (0.42)

46. Secondary Outcome: Mean Number of Paramedic Visits in Community Setting
Description: Mean number of paramedic visits in community setting for participants who were exposed to OAC and unexposed to OAC were reported in this outcome measure. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Paramedic visits
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 413083 | 265667
Paramedic visits | 28.8 (36.21) | 23.4 (38.22)

47. Secondary Outcome: Mean Number of Laboratory Tests
Description: Mean number of laboratory tests for participants who were exposed to OAC and unexposed to OAC were reported in this outcome measure. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Laboratory tests
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 369569 | 214065
Laboratory tests | 0.8 (1.31) | 0.5 (1.15)

48. Secondary Outcome: Mean Number of Outpatient Medical Procedures
Description: Mean number of outpatient medical procedures for participants who were exposed to OAC and unexposed to OAC were reported in this outcome measure. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Medical procedures
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 361232 | 221892
Medical procedures | 0.6 (0.93) | 0.5 (0.86)

49. Secondary Outcome: Mean Number of Travels Per Month
Description: Mean number of travels per month for participants who were exposed to OAC and unexposed to OAC were reported in this outcome measure. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 1
Population: Certain AF incident population included participants with a first AF diagnosis date during study period but without history of OACs delivery in the 24 months before inclusion date, with no reported events of interest (stroke, major bleeding) between inclusion and index date. Here, "Overall number of participants analyzed'' signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Travels per month
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 161349 | 127894
Travels per month | 0.3 (1.06) | 0.4 (1.32)

50. Other Pre Specified Outcome: Number of Participants According to Subgroups in OAC Exposed and Unexposed Participants
Description: The number of participants in subgroups (elderly [>=80 years], non-elderly [18 to <80 years], coronary artery disease, frail, cancer, previous stroke, high CHA₂DS₂-VASC) who were exposed to OAC and unexposed to OAC were reported in this outcome measure. Index date was the date of the first dispensation of OAC for participants exposed to OAC and for participants unexposed to OAC, index date was the date of inclusion in the study.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
Number analyzed (Participants) | 485646 | 332236
Participants
  Elderly (>=80 years) | 199562 | 170170
  Non-elderly (18 to <80 years) | 286084 | 162066
  Coronary artery disease | 86531 | 75022
  Frail | 103521 | 120900
  Active cancer | 75261 | 86281
  Previous stroke | 48610 | 32268
  High CHA2DS2-VASc | 402191 | 281168

ADVERSE EVENTS:
Time Frame: Not applicable as All-Cause Mortality, Serious, and Other [Not Including Serious] Adverse Events were not monitored/assessed
Description: Due to non-interventional nature of the study and nature of data sources, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) could not be met, hence, serious adverse events and other (non-serious adverse events) were not assessed or monitored (thus at risk appears "0"). All-cause mortality was not assessed/monitored in this study.
Arm/Group | Participants Exposed to OACs | Participants Unexposed to OACs
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publication until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (2):
  • Study Protocol (2021-12-06): https://cdn.clinicaltrials.gov/large-docs/64/NCT05838664/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-04): https://cdn.clinicaltrials.gov/large-docs/64/NCT05838664/SAP_001.pdf